CLINICAL TRIAL: NCT01765231
Title: Prophylactic Use of Entecavir for HBsAg Negative/HBcAb Positive/Hepatitis B Virus DNA Negative Patients With Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Peking University Cancer Hospital & Institute, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-2012111305
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Hepatitis B
Keywords: Lymphoma; Hepatitis B virus; Therapeutic Uses; Antiviral Agents
MeSH Terms: conditions — Hepatitis B; Lymphoma | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Entecavir prophylaxis (Experimental): Participants will initiate entecavir 0.5 mg/day orally on day 1 of the first course of antitumor therapy, and will be continued until at least 6 months after completion of antitumor therapy.
  Interventions: Drug: Entecavir prophylaxis
- Observation arm (Active Comparator): Entecavir 0.5mg daily will be prescribed for patients with hepatitis B virus reactivation.
  Interventions: Drug: Observation arm

INTERVENTIONS:
Drug: Entecavir prophylaxis — Entecavir 0.5mg daily from day 1 of antitumor therapy to at least 6 months after completing antitumor therapy
  Other Names: Baraclude
  Arms: Entecavir prophylaxis
Drug: Observation arm — Entecavir 0.5mg daily will be prescribed for patients with hepatitis B virus reactivation.
  Other Names: Therapeutic entecavir group
  Arms: Observation arm

SUMMARY:
The purpose of this study is to identify the effect of prophylactic entecavir in HBsAg Negative/HBcAb Positive/hepatitis B virus DNA Negative patients with lymphoma.

DETAILED DESCRIPTION:
The purpose of this study is to identify the effect of prophylactic entecavir in HBsAg Negative/HBcAb Positive/hepatitis B virus DNA Negative patients with lymphoma are randomized into entecavir prophylaxis group or observation group. In entecavir prophylaxis group, entecavir 0.5 mg/day orally is initiate on day 1 of the first course of antitumor therapy, and will be continued until at least 6 months after completion of antitumor therapy. In observation group, entecavir 0.5mg daily will be prescribed for patients with hepatitis B virus reactivation.

ELIGIBILITY:
Inclusion Criteria:

* treatment-naive patients with lymphoma
* HBsAg negative/HBcAb positive/hepatitis B virus DNA negative at baseline
* treated with chemotherapy and/or immunosuppressive therapy
* life expectancy of more than 3 months

Exclusion Criteria:

* younger than 18 years old
* HBsAg positive or HBcAb negative or hepatitis B virus DNA positive at baseline
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of hepatitis B virus reactivation and hepatitis B virus reactivation related hepatitis | from the beginning of anti-tumor therapy to 18 months after the last cycle of anti-tumor therapy

SECONDARY OUTCOMES:
the incidence of hepatitis B virus maintained response, the incidence of hepatitis B virus sustained response, the incidence of hepatitis B virus relapse and hepatitis B virus relapse related hepatitis | from the beginning of anti-tumor therapy to 18 months after the last cycle of anti-tumor therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (13):
- China (13):
  - Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality
  - 307 Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality
  - 309 Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Aerospace Central Hospital, Beijing, Beijing Municipality
  - Air Force General Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - First Hospital affiliated to General Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality
  - General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality